CLINICAL TRIAL: NCT03971643
Title: Open Label Exploratory Phase IIa Trial to Investigate the Safety and Efficacy of IFX-1 in Treating Patients With Pyoderma Gangrenosum (OPTIMA)
Brief Title: Exploratory Study of IFX-1 in Patients With Pyoderma Gangrenosum
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InflaRx GmbH (Industry)
Collaborators: Innovaderm Research Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFX-1-P2.7
Record Dates: First submitted 2019-05-28; First posted 2019-06-03 (Actual); Results first posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Pyoderma Gangrenosum
MeSH Terms: conditions — Pyoderma Gangrenosum | interventions — vilobelimab

STUDY DESIGN:
Intervention Model Description: IV infusions of vilobelimab diluted in sodium chloride
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- vilobelimab 800 mg Q2W (Experimental): Dose finding with a total of 15 doses of vilobelimab.
  Vilobelimab: IV infusions of vilobelimab diluted in sodium chloride.
  All patients received vilobelimab 800 mg three times during the first week (Days 1, 4, and 8).
  Starting at Day 15:
  Group 1 (N=6) continued to receive vilobelimab 800 mg every 2 weeks (Q2W), with option to increase dose from Day 57 to 1600 mg every Q2W.
  Interventions: Drug: vilobelimab
- vilobelimab 1600 mg Q2W (Experimental): Dose finding with a total of 15 doses of vilobelimab.
  Vilobelimab: IV infusions of vilobelimab diluted in sodium chloride.
  All patients received vilobelimab 800 mg three times during the first week (Days 1, 4, and 8).
  Starting at Day 15:
  Group 2 (N=6) received vilobelimab 1600 mg every 2 weeks (Q2W), with option to increase dose from Day 57 to 2400 mg every Q2W.
  Interventions: Drug: vilobelimab
- vilobelimab 2400 mg Q2W (Experimental): Dose finding with a total of 15 doses of vilobelimab.
  Vilobelimab: IV infusions of vilobelimab diluted in sodium chloride.
  All patients received vilobelimab 800 mg three times during the first week (Days 1, 4, and 8).
  Starting at Day 15:
  Group 3 (N=7) received vilobelimab 2400 mg every Q2W.
  Interventions: Drug: vilobelimab

INTERVENTIONS:
Drug: vilobelimab — IV infusions of vilobelimab diluted in sodium chloride.
  Other Names: IFX-1; CaCP29

SUMMARY:
The purpose of this study is to determine whether vilobelimab (development name: IFX-1) is safe and effective in the treatment of pyoderma gangrenosum.

DETAILED DESCRIPTION:
Neutrophilic dermatoses are a spectrum of inflammatory disorders characterized by skin lesions resulting from a neutrophil-rich inflammatory infiltrate in the absence of infection. Pyoderma gangrenosum is associated with a neutrophilic leukocytosis, which is likely to be triggered by C5a. This study is set up based on the hypothesis that vilobelimab might be able to block C5a induced pro-inflammatory effects such as neutrophil activation and cytokine generation, potentially contributing to the local skin inflammation and tissue damage.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an ulcerative form of pyoderma gangrenosum confirmed by the investigator

In addition, the subject must fulfill at least 3 of the following 6 criteria at screening:

History of

* Pathergy (ulcer occurring at the sites of trauma)
* Personal history of inflammatory bowel disease or inflammatory arthritis
* History of papule, pustule or vesicle that rapidly ulcerated

Clinical examination (or photographic evidence) of

* Peripheral erythema, undermining border, and tenderness at site of ulceration
* Multiple ulcerations (at least 1 occurring on the lower leg)
* Cribriform or "wrinkled paper" scar(s) at sites of healed ulcers

Subject has a minimum of 1 evaluable ulcer (≥2 cm2) on the lower extremity at screening

Exclusion Criteria:

* Pyoderma gangrenosum target ulcer for more than 3 years before screening
* Surgical wound debridement within the previous 2 weeks before screening
* Use of intravenous antibacterials, antivirals, anti-fungals, or anti-parasitic agents within 30 days before screening
* Any drug treatment for pyoderma gangrenosum including corticosteroids (>10 mg), intralesional steroids, cyclosporine A, biologicals and immunosuppressives (with the exception of antibiotics for wound superinfection) used within a time of 5 half-lives of the drug before screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Niels C. Riedemann, M.D., Ph.D., Study Director — InflaRx GmbH
Locations (10):
- United States (7):
  - InflaRx Site #07, Sacramento, California
  - InflaRx Site #08, Miami, Florida
  - InflaRx Site #03, Tampa, Florida
  - InflaRx Site #10, St Louis, Missouri
  - InflaRx Site #05, Columbus, Ohio
  - InflaRx Site #12, Hershey, Pennsylvania
  - InflaRx Site #09, Pittsburgh, Pennsylvania
- InflaRx Site #01, Richmond Hill, Ontario, Canada
- Poland (2):
  - InflaRx Site #21, Rzeszów
  - InflaRx Site #20, Wroclaw

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vilobelimab 800 mg Q2W: Group 1 (N=6) continued to receive vilobelimab 800 mg every 2 weeks (Q2W), with option to increase dose from Day 57 to 1600 mg every Q2W.
- Vilobelimab 1600 mg Q2W: Group 2 (N=6) received vilobelimab 1600 mg every 2 weeks (Q2W), with option to increase dose from Day 57 to 2400 mg every Q2W.
- Vilobelimab 2400 mg Q2W: Group 3 (N=7) received vilobelimab 2400 mg every 2 weeks (Q2W).
Period: Overall Study
Arm/Group | Vilobelimab 800 mg Q2W | Vilobelimab 1600 mg Q2W | Vilobelimab 2400 mg Q2W
Started | 6 | 6 | 7
Completed Until Day 99 (Evaluable) | 6 | 4 | 7
Completed | 1 | 3 | 6
Not Completed | 5 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vilobelimab 800 mg Q2W | Vilobelimab 1600 mg Q2W | Vilobelimab 2400 mg Q2W | Total
Number analyzed (Participants) | 6 | 6 | 7 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (11.41) | 60.5 (12.36) | 43.0 (15.00) | 53.7 (14.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 10
  Male | 2 | 3 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 6 | 6 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 6 | 4 | 7 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Baseline Disease Characteristic: Duration of pyoderma gangrenosum [Mean (Standard Deviation); unit: years] | 1.7 (1.86) | 5.7 (9.54) | 3.4 (6.05) | 3.6 (6.41)
Baseline Disease Characteristic: Wound area at baseline [Mean (Standard Deviation); unit: area [mm²]] — Population: For two patients the measurements could not be obtained because photos were not taken correctly.
  area [mm²]
    number analyzed (Participants) | 5 | 5 | 7 | 17
    (all) | 1692.374 (1391.4307) | 7898.952 (5844.5941) | 1827.553 (1901.2830) | 3573.500 (4320.3723)

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Adverse Events (TEAEs), Related TEAEs, Serious TEAEs, and Adverse Events of Special Interest (AESIs)
Description: Number of patients with treatment-emergent adverse events (TEAEs), related TEAEs, serious TEAEs, and adverse events of special interest (AESIs)
  TEAEs are defined as adverse events that start at or after the first administration of study drug.
  Related TEAEs are defined as all TEAEs considered by the investigator to have at least a 'possible' relationship with the study drug.
  AESIs are defined as infusion-related reactions, including acute and delayed hypersensitivity and anaphylactic reactions during or after infusion; Meningitis; Meningococcal septicaemia; Invasive infection.
  As adverse events will be reported in details in the safety section, no separate reporting on System Organ Class (SOC) or Preferred Term (PT) level etc. is done here.
Time Frame: From treatment start until end of study (including observational visits), an average of 249 days
Population: Safety set
Measure: Count of Participants; unit: Participants
Groups:
- Vilobelimab 800 mg Q2W: Group 1 (N=6) continued to receive vilobelimab 800 mg every 2 weeks (Q2W),with option to increase dose from Day 57 to 1600 mg every Q2W.
Arm/Group | Vilobelimab 800 mg Q2W | Vilobelimab 1600 mg Q2W | Vilobelimab 2400 mg Q2W
Number analyzed (Participants) | 6 | 6 | 7
Participants
  Treatment-emergent adverse events (TEAEs) | 6 | 4 | 5
  Related TEAEs | 0 | 2 | 2
  Serious TEAEs | 1 | 1 | 2
  Adverse events of special interest (AESIs) as identified by investigator | 0 | 1 | 1
  Adverse events of special interest (AESIs) as identified by sponsor | 2 | 1 | 2

2. Secondary Outcome: Number of Patients With Physician's Global Assessment (PGA) Score ≤3 (Investigator Assessment)
Description: Efficacy endpoint: Proportion of patients with a clinical response, defined as Physician's Global Assessment (PGA) score ≤3 of target ulcer at Visit V4, V6, V10 and V16 (End of Treatment [EOT]) (SAF).
  PGA values: 0 = Completely clear, 1 = Almost clear, 2 =Marked improvement, 3 = Moderate improvement, 4 = Slight improvement, 5 = No change from baseline, 6 = Worse
Time Frame: From treatment start until V16 (Day 189)
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Vilobelimab 800 mg Q2W | Vilobelimab 1600 mg Q2W | Vilobelimab 2400 mg Q2W
Number analyzed (Participants) | 6 | 6 | 7
Participants
  V4 | 2 | 0 | 0
  V6: number analyzed (Participants) | 6 | 4 | 7
  V6 | 1 | 1 | 3
  V10: number analyzed (Participants) | 6 | 4 | 6
  V10 | 3 | 1 | 5
  V16: number analyzed (Participants) | 1 | 3 | 6
  V16 | 0 | 1 | 5

3. Secondary Outcome: Time to Complete Closure of Pyoderma Gangrenosum Target Ulcer (Investigator Assessment) [Days]
Description: Efficacy endpoint: Kaplan-Meier analysis of time to first clinical remission (complete closure of target ulcer) defined as PGA score of ≤ 1,
  PGA values: 0 = Completely clear, 1 = Almost clear, 2 =Marked improvement, 3 = Moderate improvement, 4 = Slight improvement, 5 = No change from baseline, 6 = Worse
Time Frame: From treatment start until end of study (including observational visits), an average of 249 days
Population: Safety Set
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Vilobelimab 800 mg Q2W | Vilobelimab 1600 mg Q2W | Vilobelimab 2400 mg Q2W
Number analyzed (Participants) | 6 | 6 | 7
days | NA [62 to NA] — Not available as values were not calculable due to low number of responders | NA [NA to NA] — Not available as values were not calculable due to low number of responders | 126 [77 to 197]

4. Secondary Outcome: Percentage Change in Wound Healing (Wound Area) by Photographic Assessment
Description: Efficacy endpoint: Percentage change in wound area [percent change] of target ulcer by photographic assessment between Visits V1 and V4, between Visits V1 and V6, between Visits V1 and V16, between Visits V6 and V10, between Visits V10 and V16.
Time Frame: From treatment start until V16 (Day 189)
Population: Safety Set
  Only patients with an available wound area measurement at both relevant visits are included in the respective analysis. Wound area for single visits was missing because images were not taken correctly and the measurements could not be obtained or patients discontinued the study prior to the relevant visit.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Vilobelimab 1600 mg Q2W: Group 2 (N=6) received Ivilobelimab 1600 mg every 2 weeks (Q2W), with option to increase dose from Day 57 to 2400 mg every Q2W.
Arm/Group | Vilobelimab 800 mg Q2W | Vilobelimab 1600 mg Q2W | Vilobelimab 2400 mg Q2W
Number analyzed (Participants) | 6 | 6 | 7
percent change
  V1-V4: number analyzed (Participants) | 5 | 5 | 7
  V1-V4 | -13.612 (41.7862) | 16.099 (15.0992) | -12.620 (31.9371)
  V1-V6: number analyzed (Participants) | 5 | 3 | 7
  V1-V6 | -4.130 (74.1725) | -8.413 (47.5261) | -34.153 (53.3455)
  V1-V16: number analyzed (Participants) | 1 | 2 | 6
  V1-V16 | 234.068 | -57.538 (60.0506) | -90.918 (16.2280)
  V6-V10: number analyzed (Participants) | 6 | 4 | 6
  V6-V10 | -22.803 (52.8937) | -16.198 (58.8229) | -63.059 (50.1507)
  V10-V16: number analyzed (Participants) | 1 | 2 | 3
  V10-V16 | 61.451 | 8.644 (5.2038) | -51.141 (69.4133)

5. Secondary Outcome: Percentage Change in Wound Healing (Wound Volume) by Photographic Assessment
Description: Efficacy endpoint: Percentage change in wound volume [percent change] of target ulcer by photographic assessment between Visits V1 and V4, between Visits V1 and V6, between Visits V1 and V16, between Visits V6 and V10, between Visits V10 and V16.
Time Frame: From treatment start until V16 (Day 189)
Population: Safety Set
  Only patients with an available wound volume measurement at both relevant visits are included in the respective analysis. Wound volume for single visits was missing because images were not taken correctly and the measurements could not be obtained or patients discontinued the study prior to the relevant visit. Additionally, sometimes the pictures allowed to measure the wound area, but not the volume as several pictures had to be taken to estimate the volume adequately.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vilobelimab 800 mg Q2W | Vilobelimab 1600 mg Q2W | Vilobelimab 2400 mg Q2W
Number analyzed (Participants) | 6 | 6 | 7
percent change
  V1-V4: number analyzed (Participants) | 5 | 1 | 4
  V1-V4 | -19.733 (53.4282) | 74.918 | -36.328 (32.3445)
  V1-V6: number analyzed (Participants) | 4 | 0 | 3
  V1-V6 | -17.300 (90.9283) |  | -58.959 (46.7969)
  V1-V16: number analyzed (Participants) | 1 | 0 | 5
  V1-V16 | 786.937 |  | -92.639 (15.6580)
  V6-V10: number analyzed (Participants) | 4 | 1 | 3
  V6-V10 | -38.033 (82.8031) | -100.000 | -82.525 (30.2680)
  V10-V16: number analyzed (Participants) | 1 | 0 | 3
  V10-V16 | 150.857 |  | 4.167 (177.7658)

6. Secondary Outcome: Rate of Change Per Day in Area of Target Ulcer by Photographic Assessment From V1 to V16
Description: Efficacy endpoint: Rate of change per day in area of target ulcer [mm²/day] between Visits V1 and V16 (photographic assessment)
Time Frame: From treatment start until V16 (Day 189)
Population: Safety Set
  Only patients with an available wound area measurement at both relevant visits (V1 and V16) are included in this analysis. Wound area for single visits was missing because images were not taken correctly and the measurements could not be obtained or patients discontinued the study prior to the relevant visit.
Measure: Mean (Standard Deviation); unit: mm²/day
Arm/Group | Vilobelimab 800 mg Q2W | Vilobelimab 1600 mg Q2W | Vilobelimab 2400 mg Q2W
Number analyzed (Participants) | 1 | 2 | 6
mm²/day | 15.14 | -12.04 (9.638) | -9.58 (10.751)

7. Secondary Outcome: Number of Patients With ≥ 50% Decrease in Area of Target Ulcer by Photographic Assessment at V16
Description: Efficacy endpoint: Number of patients with a decrease in area of target ulcer of ≥ 50% by photographic assessment at Visit V16 (EOT) compared to Baseline
Time Frame: From treatment start until V16 (Day 189)
Population: Safety Set
  Only patients with an available wound area measurement at baseline and V16 are included in this analysis. Wound area for single visits was missing because images were not taken correctly and the measurements could not be obtained or patients discontinued the study prior to the relevant visit.
Measure: Count of Participants; unit: Participants
Groups:
- Vilobelimab 1600 mg Q2W: Group 2 (N=6) received vilobelimab 1600 mg every 2 weeks (Q2W), with option to increase dose from Day 57 to 2400 mg every two week (Q2W).
Arm/Group | Vilobelimab 800 mg Q2W | Vilobelimab 1600 mg Q2W | Vilobelimab 2400 mg Q2W
Number analyzed (Participants) | 1 | 2 | 6
Participants | 0 | 1 | 6

8. Secondary Outcome: Number of Patients With 100% Decrease in Area of Target Ulcer at V16
Description: Efficacy endpoint: Number of patients with a decrease in area of target ulcer of 100% at Visit V16 (EOT) compared to Baseline (remission) (photographic assessment)
Time Frame: From treatment start until V16 (Day 189)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Vilobelimab 800 mg Q2W | Vilobelimab 1600 mg Q2W | Vilobelimab 2400 mg Q2W
Number analyzed (Participants) | 1 | 2 | 6
Participants | 0 | 1 | 2

9. Secondary Outcome: Degree of Erythema of the Target Ulcer at V4, V6, V10 and V16
Description: Efficacy endpoint: Degree of erythema of the target ulcer at Visit V4, V6, V10 and V16 (EOT) (investigator assessment)
Time Frame: From treatment start until V16 (Day 189)
Population: Safety set
Measure: Count of Participants; unit: Participants
Arm/Group | Vilobelimab 800 mg Q2W | Vilobelimab 1600 mg Q2W | Vilobelimab 2400 mg Q2W
Number analyzed (Participants) | 6 | 6 | 7
Participants
  V4: None (0) | 0 | 0 | 0
  V4: Slight (1) | 0 | 0 | 0
  V4: Moderate (2) | 2 | 2 | 1
  V4: Severe (3) | 3 | 3 | 4
  V4: Very severe (4) | 1 | 1 | 2
  V6: number analyzed (Participants) | 6 | 4 | 7
  V6: None (0) | 1 | 0 | 0
  V6: Slight (1) | 0 | 0 | 1
  V6: Moderate (2) | 2 | 2 | 2
  V6: Severe (3) | 2 | 2 | 3
  V6: Very severe (4) | 1 | 0 | 1
  V10: number analyzed (Participants) | 6 | 4 | 6
  V10: None (0) | 1 | 0 | 0
  V10: Slight (1) | 0 | 1 | 3
  V10: Moderate (2) | 3 | 1 | 1
  V10: Severe (3) | 2 | 2 | 2
  V10: Very severe (4) | 0 | 0 | 0
  V16: number analyzed (Participants) | 1 | 3 | 6
  V16: None (0) | 0 | 1 | 0
  V16: Slight (1) | 0 | 1 | 5
  V16: Moderate (2) | 0 | 0 | 1
  V16: Severe (3) | 1 | 1 | 0
  V16: Very severe (4) | 0 | 0 | 0

10. Secondary Outcome: Border Elevation of the Target Ulcer at Visits V4, V6, V10 and V16
Description: Efficacy endpoint: Border elevation of the target ulcer at visits V4, V6, V10 and V16 (EOT) (investigator assessment)
Time Frame: From treatment start until V16 (Day 189)
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Vilobelimab 800 mg Q2W | Vilobelimab 1600 mg Q2W | Vilobelimab 2400 mg Q2W
Number analyzed (Participants) | 6 | 6 | 7
Participants
  V4: None (0) | 0 | 0 | 0
  V4: Slight (1) | 2 | 0 | 0
  V4: Moderate (2) | 1 | 5 | 4
  V4: Severe (3) | 3 | 0 | 3
  V4: Very severe (4) | 0 | 1 | 0
  V6: number analyzed (Participants) | 6 | 4 | 7
  V6: None (0) | 2 | 0 | 1
  V6: Slight (1) | 1 | 0 | 1
  V6: Moderate (2) | 2 | 3 | 4
  V6: Severe (3) | 1 | 1 | 1
  V6: Very severe (4) | 0 | 0 | 0
  V10: number analyzed (Participants) | 6 | 4 | 6
  V10: None (0) | 1 | 0 | 0
  V10: Slight (1) | 2 | 1 | 6
  V10: Moderate (2) | 3 | 3 | 0
  V10: Severe (3) | 0 | 0 | 0
  V10: Very severe (4) | 0 | 0 | 0
  V16: number analyzed (Participants) | 1 | 3 | 6
  V16: None (0) | 0 | 1 | 1
  V16: Slight (1) | 0 | 1 | 4
  V16: Moderate (2) | 1 | 1 | 1
  V16: Severe (3) | 0 | 0 | 0
  V16: Very severe (4) | 0 | 0 | 0

11. Secondary Outcome: Percentage Change in Pain by Numeric Rating Scale (NRS) at Visits V4, V6, V10 and V16
Description: Efficacy endpoint: Percentage change from Baseline in pain assessed by Numeric Rating Scale (NRS) [percent change] at visits V4, V6, V10 and V16 (EOT) Mean (SD)
  The NRS is an 11-point scale (from 0 represent no pain to 10 representing the worst pain the subject can imagine).
Time Frame: From treatment start until V16 (Day 189)
Population: Safety set
  Only patients with an available NRS at both relevant visits are included in the respective analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vilobelimab 800 mg Q2W | Vilobelimab 1600 mg Q2W | Vilobelimab 2400 mg Q2W
Number analyzed (Participants) | 6 | 6 | 7
percent change
  V1-V4: number analyzed (Participants) | 5 | 5 | 7
  V1-V4 | -41.6 (31.29) | 10.6 (19.88) | -41.4 (33.77)
  V1-V6: number analyzed (Participants) | 5 | 4 | 7
  V1-V6 | -43.3 (16.43) | 1.7 (22.19) | -45.0 (45.23)
  V1-V10: number analyzed (Participants) | 4 | 4 | 6
  V1-V10 | -64.3 (32.55) | 32.5 (89.87) | -72.2 (32.07)
  V1-V16: number analyzed (Participants) | 1 | 3 | 6
  V1-V16 | -22.2 | 5.6 (141.75) | -51.6 (33.89)

12. Secondary Outcome: Percentage Change in Life Quality by DLQI at Visits V4, V6, V10, and V16
Description: Efficacy endpoint: Percentage change from Baseline in Dermatology Life Quality Index (DLQI) [percent change] at visits V4, V6, V10, and V16 (EOT)
  The DLQI comprises 10 questions with single scores 0 (No effect on patient's life) to 3 (large effect on patient's life). The DLQI total score is calculated by summing up the score of each question resulting in a minimum of 0 (best) and a maximum of 30 (worst).
Time Frame: From treatment start until V16 (Day 189)
Population: Safety set
  Only patients with an available DLQI at both relevant visits are included in the respective analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Vilobelimab 800 mg Q2W | Vilobelimab 1600 mg Q2W | Vilobelimab 2400 mg Q2W
Number analyzed (Participants) | 6 | 6 | 7
percent change
  V1-V4 | -29.9 (22.75) | -3.8 (51.05) | -33.1 (28.61)
  V1-V6: number analyzed (Participants) | 6 | 4 | 7
  V1-V6 | -31.4 (20.29) | -33.2 (29.68) | -24.7 (34.30)
  V1-V10: number analyzed (Participants) | 6 | 4 | 6
  V1-V10 | -50.0 (28.01) | -33.9 (31.26) | -43.1 (28.17)
  V1-V16: number analyzed (Participants) | 1 | 3 | 6
  V1-V16 | 4.5 | -2 (56.07) | -50.8 (45.10)

ADVERSE EVENTS:
Time Frame: From treatment start until end of study (including observational visits), an average of 249 days
Arm/Group | Vilobelimab 800 mg Q2W | Vilobelimab 1600 mg Q2W | Vilobelimab 2400 mg Q2W
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 2/7
Other Adverse Events (participants affected / at risk) | 6/6 | 3/6 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vilobelimab 800 mg Q2W (N=6) | Vilobelimab 1600 mg Q2W (N=6) | Vilobelimab 2400 mg Q2W (N=7)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Superinfection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vilobelimab 800 mg Q2W (N=6) | Vilobelimab 1600 mg Q2W (N=6) | Vilobelimab 2400 mg Q2W (N=7)
Wound infection (Infections and infestations) | 2 (3) | 1 (1) | 0 (0)
Wound infection pseudomonas (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Lichen planus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Traumatic haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Glossitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Superficial vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results of the Study conducted at the Study Site shall not be made before the first multi-site publication by Sponsor occured within 18 months

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT03971643/Prot_SAP_002.pdf
  • Informed Consent Form (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT03971643/ICF_003.pdf